CLINICAL TRIAL: NCT06134375
Title: Novel Targeting of the Microenvironment to Decrease Metastatic Recurrence of High-Risk TNBC: A Randomized Phase II Study of Tetrathiomolybdate (TM) Plus Capecitabine in Patients With Breast Cancer at High Risk of Recurrence
Brief Title: A Study of Tetrathiomolybdate (TM) Plus Capecitabine
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Linda.T.Vahdat, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY02001837; R01CA290013 (NIH); CDMRP-eBRAP BC240345 (Other Grant/Funding Number: Department of Defense); 22VAH837 (Other: Dartmouth Hitchcock); NCI-2025-05879 (Other: NCI ID)
Record Dates: First submitted 2023-10-03; First posted 2023-11-18 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Triple Negative Breast Cancer; Residual Disease
Keywords: Triple Negative Breast cancer; Residual Disease
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Neoplasm, Residual | interventions — tetrathiomolybdate; Capecitabine; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Phase 1 portion is single group. Phase 2 portion is parallel.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- TM and Capecitabine with or without Pembrolizumab (Experimental): Tetrathiomolybdate (TM) and Capecitabine +/- Pembrolizumab will be administered concurrently for 6 months, TM will continue for 2.5 more years (total duration of TM treatment is 3 years)
  Interventions: Drug: Tetrathiomolybdate; Drug: Capecitabine; Drug: Pembrolizumab
- Capecitabine with or without Pembrolizumab (Active Comparator): Capecitabine +/- Pembrolizumab will be administered for 6 months (participants will remain on study for 2.5 more years).
  Interventions: Drug: Capecitabine; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Tetrathiomolybdate — Tetrathiomolybdate (TM): Ammonium tetrathiomolybdate (TM), an oral copper lowering agent, has been established as safe in patients with Wilson's disease and advanced cancer. TM forms stable copper-molybdenum clusters sequestering copper and thereby limiting its availability, for the proper functioning of angiogenic factors, including secreted metalloenzymes. TM inhibits several copper containing enzymes including ceruloplasmin, cytochrome oxidase, tyrosinase and downregulates cytokines such as MMP9 and VEGF as well as transcription factors such as NF-kB. Both pre-clinical and clinical data suggest that TM may effectively reduce both overt and sub-clinical tumor load by both targeting the metastases initiating stem cell component of primary tumors inactivating Complex IV, shifting oxphos to glycolysis and through stromal remodeling.
  Other Names: TM
  Arms: TM and Capecitabine with or without Pembrolizumab
Drug: Capecitabine — 1000mg/m2 twice daily, Days 1-14 Q21days for 6 months
  Other Names: Xeloda
Drug: Pembrolizumab — If pembrolizumab was administered in the neoadjuvant setting and the oncology team chooses to continue in the adjuvant setting, standard doses will be used (200 mg IV Q3weeks or 400 mg IV Q6 weeks for one year total as per package insert)
  Other Names: Keytruda

SUMMARY:
There are two parts to this study. It is a phase 1b followed by a randomized phase 2 study to assess whether adding 3 years of adjuvant tetrathiomolybdate (TM) to standard 6 months treatment of adjuvant capecitabine and pembrolizumab in high risk for relapse triple negative breast cancer.

In the phase 1b part of the study, TM is added to adjuvant capecitabine and pembrolizumab in high risk for relapse triple negative breast cancer (RCB 2, 3, risk for relapse >60% at 5 years) after completion of neoadjuvant chemo-immunotherapy and surgery to establish the safety of the combination. This will be followed by a randomized phase 2 clinical trial of adjuvant TM and capecitabine vs capecitabine alone.

If pembrolizumab was administered in the neoadjuvant setting, it may be continued in the adjuvant setting per investigator discretion.

DETAILED DESCRIPTION:
Scientific Rationale for the study design: Copper depletion is designed to be a complement to standard therapy to overcome resistance mechanisms hence it would be optimal to combine it with standard adjuvant therapy which at the current time is capecitabine and pembrolizumab.

Study Design:

Phase 1b: Patients with triple negative breast cancer who have completed standard neoadjuvant therapy (chemotherapy + pembrolizumab) and who have residual disease at RCB 2, 3 will start adjuvant therapy with standard dose capecitabine, standard dose pembrolizumab and tetrathiomolybdate (TM). Patients must have received neoadjuvant immunotherapy (pembrolizumab) and wish to continue adjuvant immunotherapy for at least one cycle on trial. The capecitabine will be for 6 months with concurrent TM and TM will continue for an additional 2.5 years (for a total of 3 years of treatment). Patients must stay on immunotherapy for at least the first cycle of the study and subsequently as per physician's choice.

This phase of the study is designed to assess safety of TM with capecitabine + immunotherapy (pembrolizumab) as adjuvant therapy for TNBC.

With a standard 3+3 design, the maximum possible total number of patients is 18.

Randomized Phase 2: Patients with triple negative breast cancer who have completed standard neoadjuvant therapy (chemotherapy +/- pembrolizumab) and who have residual disease at RCB 2, 3 will start adjuvant therapy with standard dose capecitabine or capecitabine and tetrathiomolybdate (TM). If they received neoadjuvant pembrolizumab and wish to continue adjuvant immunotherapy, they may continue. The capecitabine will be for 6 months with concurrent TM and TM will continue for an additional 2.5 years (for a total of 3 years of treatment). If they elect to continue immunotherapy, then they should complete one year total or as per physician's choice.

Patients will be randomized with a 1:1 allocation ratio between the two treatment arms.

There will be at most 186 patients accrued to account for 10% loss to follow-up over the course of the approximately 5-year study period.

Study Treatment:

Phase 1b:

• Induction Phase TM dose: as per dose escalation nomogram. Dose Level 1 is 140 mg a day (TM 100 mg + 40 mg QHS) Ceruloplasmin (Cp) target: Will be done at local lab. The Cp target goal is to be 1-6 mg/dL below the lower limit of normal for the reference lab (see Section 7.1).

Capecitabine Dose: 1000 mg per square meter of body-surface area, twice per day, on days 1 to 14 every 3 weeks.

Pembrolizumab: Standard doses will be used (200 mg IV Q3 weeks or 400 mg IV Q6 weeks

• Maintenance Phase TM dose: as per dose escalation nomogram Dose Level 1 is 100 mg a day (TM 100 mg daily) Cp target: Will be done at local lab. Goal is to be 1-6 mg/dL below the lower limit of normal for the reference lab (see Section 7.1). TM dosed according to Cp level and ANC in 20mg TM capsule increments.

Capecitabine Dose: 1000 mg per square meter of body-surface area, twice per day, on days 1 to 14 every 3 weeks for a total of 6 months Pembrolizumab: Standard doses will be used (200 mg IV Q3 weeks or 400 mg IV Q6 weeks for one year total as per package insert or per physician's choice).

Study Duration: TM and capecitabine and pembrolizumab will be administered concurrently for 6 months, and the TM will continue for an additional 2.5 years (total duration of TM treatment is 3 years).

If no DLT is observed at dose level +2 then that is the dose that will proceed to the randomized phase 2 portion of the study.

Randomized Phase 2:

* Randomization: Patients will be randomized 1:1 to the combination of Capecitabine and TM vs. Capecitabine. If pembrolizumab was administered in the neoadjuvant setting and the oncology team chooses to continue in the adjuvant setting, standard doses will be used (200 mg IV Q3weeks or 400 mg IV Q6 weeks for one year total as per package insert or per physician's choice)
* Induction Phase TM dose: Will be determined in phase 1b part of this study. If no DLT noted at dose level 2, then will proceed with TM dose 180 mg a day (TM 100 mg qAM + 80 mg QHS) Cp target: Will be done at local lab. Goal is to be 1-6 mg/dL below the lower limit of normal for the reference lab (see Section 7.1) Capecitabine Dose: 1000 mg per square meter of body-surface area, twice per day, on days 1 to 14 every 3 weeks for a total of 6 months Pembrolizumab: optional as per physician's choice. Standard doses will be used (200 mg IV Q3weeks or 400 mg IV Q6 weeks for one year total per package insert or per physician's choice
* Maintenance Phase TM dose: Will be determined in phase 1b part of this study. If no DLT noted at dose level 2, then will proceed with TM dose 100 mg a day (TM 100 mg QD) Cp target: Will be done at local lab. Goal is to be 1-6 mg/dL below the lower limit of normal for the reference lab (see Section 7.1). TM dosed according to Cp level and ANC in 20mg TM capsule increments.

Capecitabine Dose: 1000 mg per square meter of body-surface area, twice per day, on days 1 to 14 every 3 weeks for a total of 6 months Pembrolizumab: optional as per physician's choice. Standard doses will be used (200 mg IV Q3weeks or 400 mg IV Q6 weeks for one year total per package insert or per physician's choice.

Study Duration: TM and capecitabine will be administered concurrently for 6 months, and the TM will continue for an additional 2.5 years (total duration of TM treatment is 3 years). Pembrolizumab is optional and should be administered according to standard guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed breast malignancy that is Triple negative tumors as defined as ER and PR <1% and HER2 negative as per ASCO/CAP guidelines
2. The patient must have completed standard neoadjuvant chemotherapy which constitutes at least 6 cycles of chemotherapy.
3. Phase Ib: Patients must have residual invasive carcinoma, at minimum in one of the following capacities: (1) node positive disease after treatment without residual invasive carcinoma in the breast; (2) RCB 2 or RCB 3 MDAH Calculator; Standard therapy consists of the following: (1) Local therapy: (a) Lumpectomy or mastectomy to negative margins. (b) Sentinel lymph node biopsy or axillary node dissection; (c) Radiation therapy to breast if patient received a lumpectomy and per investigator choice if considering chest wall/extended field RT. (2) Systemic therapy: Prior chemotherapy is required for patients entered on the trial. Neoadjuvant treatment should consist of the following standard therapy: Anthracycline and taxane-based therapy (i.e. AC->T, AC->Tcarbo, Keynote 522 regimen) or a non-anthracycline based chemo and immunotherapy regimen (NeoPACT). Patients must have received neoadjuvant Pembrolizumab for the phase Ib only and plan to continue it in the adjuvant setting for at least the first cycle of treatment.

   Randomized Phase 2: Patients must have residual invasive carcinoma, at minimum in one of the following capacities: (1) node positive disease after treatment without residual invasive carcinoma in the breast; (2) RCB 2 or RCB 3 MDAH Calculator; Standard therapy consists of the following: (1) Local therapy: (a) Lumpectomy or mastectomy to negative margins. (b) Sentinel lymph node biopsy or axillary node dissection; (c) Radiation therapy to breast if patient received a lumpectomy and per investigator choice if considering chest wall/extended field RT. (2) Systemic therapy: Prior chemotherapy is required for patients entered on the trial. Neoadjuvant treatment should consist of the following standard therapy: Anthracycline and taxane-based therapy (i.e. AC->T, AC->Tcarbo, Keynote 522 regimen) or a non-anthracycline based chemo and immunotherapy regimen (NeoPACT). Pembrolizumab is allowed. Patients will be stratified by: (1) Treatment (chemotherapy vs chemotherapy + immunotherapy); (2) Age (Age ≤ 40 yrs vs > 40 yrs); and (3) RCB 2 vs RCB 3. These important stratification factors represent variables that are known to affect outcome for patients with TNBC.
4. At least two weeks must have elapsed from last chemotherapy or radiation therapy. At least 4 weeks must have elapsed from most recent surgery.
5. No clinical or radiologic evidence of disease after surgery and/or systemic treatment (by CT scan of chest, abdomen and pelvis and bone scan or PET scan prior to enrollment).
6. Previous treatment with capecitabine is not allowed.
7. Because no dosing or adverse event data are currently available on the use of TM in patients <18 years of age, children are excluded from this study.
8. KPS 90 or 100.
9. Life expectancy of greater than 3 months.
10. Patients must have normal organ and marrow function as defined below:

    * hemoglobin >10mg/dL
    * absolute neutrophil count >1,500/ µL
    * platelets >100,000/µL
    * total bilirubin <1.5 x normal institutional limits
    * AST (SGOT)/ALT (SGPT) <1.5 X institutional upper limit of normal
11. Antiresorptive therapy and denosumab may be administered.
12. Patients must be on stable medical therapy for at least 2 weeks if they are being treated medically for their chemotherapy induced peripheral neuropathy.
13. The effects of TM on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
14. Ability to understand and the willingness to sign a written informed consent document.
15. Normal B12 levels.

Exclusion Criteria:

1. Patients who have had chemotherapy or radiotherapy within 2 weeks prior to entering the study. Patients who have had surgery within 4 weeks.
2. Patients who have received capecitabine or who are on warfarin
3. Patients who had their final breast surgery more than 12 weeks prior to study start.
4. Phase Ib: patients who have not received neoadjuvant immunotherapy and/or do not plan to continue treatment with immunotherapy for at least the first cycle of study treatment.
5. Objective evidence of breast cancer.
6. Metastatic disease
7. Carcinomatous meningitis or active parenchymal brain metastases.
8. Estimated creatinine clearance < 60 ml/min
9. History of allergic reactions attributed to compounds of similar chemical or biologic composition to TM or capecitabine.
10. Pregnant women are excluded from this study because TM has the potential to have teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with TM, breastfeeding should be discontinued if the mother is treated with TM.
11. Because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, HIV-positive patients receiving combination anti- retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with TM.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2031-06-26 (Estimated); Study Completion 2036-06-26 (Estimated)

PRIMARY OUTCOMES:
Phase 1b: To establish the safety of the combination of adjuvant tetrathiomolybdate with capecitabine and pembrolizumab by the number of dose limiting toxicities | 3 years
  To establish the safety of the combination of adjuvant tetrathiomolybdate with capecitabine and pembrolizumab administered to patients with triple negative breast cancer after completion of neoadjuvant chemotherapy and with a non-pCR (RCB 2, 3) after standard surgery. The safe dose is defined as the dose level at which no more than 1 out of 6 patients has a DLT on Cycle 1. A dose limiting toxicity (DLT) is defined as a grade 3 hematologic toxicity or non-hematologic toxicity excluding hand foot syndrome, mucositis, or diarrhea. The DLT window is 4 weeks. All toxicities will be summarized.
Phase 2: Distant relapse-free survival (DRFS) between TM and capecitabine versus capecitabine as measured with the STEEP system | 10 years
  The primary endpoint of this study is distant relapse-free survival (DRFS) between TM and capecitabine versus capecitabine. The continued use of adjuvant immunotherapy with pembrolizumab is left to investigator choice. DRFS is defined in accordance with the STEEP system. This definition of DRFS, includes the following as events: distant recurrence, death from breast cancer, death from non-breast cancer or unknown causes, or any second primary invasive cancer. DRFS will be compared by arm in each of the two RCB groups separately using time-to-event analytic methods such as the log-rank test and Cox regression.

SECONDARY OUTCOMES:
Phase 1b: Distant Relapse free survival (DRFS) between TM, capecitabine and pembrolizumab versus capecitabine and pembrolizumab as measured with the STEEP system | 3 years
  Distant Relapse free survival (DRFS) between TM, capecitabine and pembrolizumab versus capecitabine and pembrolizumab. DRFS is defined in accordance with the STEEP system. This definition of DRFS, includes the following as events: distant recurrence, death from breast cancer, death from non-breast cancer or unknown causes, or any second primary invasive cancer. This will be analyzed descriptively due to small sample sizes and possibly different dose levels.
Phase 1b: Plasma concentrations of capecitabine, pembrolizumab and TM will be performed in a sub cohort of at least nine patients enrolled in the phase 1b part of this study | 3 years
  Pharmacokinetics of capecitabine, pembrolizumab and TM. Capecitabine and 5 fluoro-uracil will be measured in plasma and 5FU intracellular nucleotides will be measured in PBMCs. Plasma pembrolizumab concentrations will be measured using the commercially available ELISA assay.
Phase 2: Overall Survival compared by arm in each of the two RCB groups separately | 10 years
  Overall survival (OS) between the two arms via the Kaplan-Meier method
Phase 2: invasive disease-free survival compared by arm in each of the two RCB groups separately | 10 years
  Invasive disease-free survival (iDFS) between the two arms via the Kaplan-Meier method
Phase 2: Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 comparing capecitabine and tetrathiomolybdate +/- pembrolizumab versus capecitabine alone +/- pembrolizumab | 5 years
  Treatment-related adverse events comparing capecitabine and tetrathiomolybdate +/- pembrolizumab versus capecitabine alone +/- pembrolizumab. Safety will be described by calculating the frequencies and 95% confidence intervals for each adverse event, with the maximum grade per toxicity serving as the patient-specific summary measure. Safety in terms on adverse events will be described over the entire time period, in addition to specific time periods (after 1 year, 2 and 3 years after the start of therapy) to evaluate late onset adverse events.
Phase 2: Survival in patients that complete at least 6 months of treatment | 10 years
  Overall survival (OS) and invasive disease-free survival (iDFS) in patients that complete at least 6 months of TM and capecitabine therapy versus capecitabine alone (+/- pembrolizumab for each arm) (enough time to be copper depleted) via the Kaplan-Meier method
Phase 2: Effect of copper depletion on serial blood-based biomarkers | 5 years
  Effect of copper depletion on serial blood-based biomarkers including: VEGFR2+ EPCs, LOXL-2, ctDNA, other biomarkers in process of validation by correlation coefficients
Phase 2: Patient-reported quality of life measurements to assess whether the addition of TM to capecitabine impacts health-related quality of life and differ between arms over time | 5 years
  Patient-reported quality of life (PROs) including: oral, gastrointestinal, cutaneous, neurological, and treatment-related symptoms will be assessed every 16 weeks in both arms through surveys. The questionnaire uses a 5-point Likert scale to assess severity with a scale from none, never, not at all, etc. to very much, constantly, very severe, etc. or yes and no. Separate mixed linear models will be conducted for each symptom to compare the average difference between the randomized arms.
Phase 2: Plasma concentrations of capecitabine, pembrolizumab and TM will be performed in a sub cohort of patients enrolled in the randomized phase 2 part of this study | 5 years
  Based on the phase 1b pharmacokinetics analyses, a population pharmacokinetic sampling schema will be developed for a sub cohort (the number of participants will be determined based on the phase 1b results) in the randomized phase 2 part of the study. Pharmacokinetics of capecitabine, pembrolizumab and TM. Capecitabine and 5 fluoro-uracil will be measured in plasma and 5FU intracellular nucleotides will be measured in PBMCs. Plasma pembrolizumab concentrations will be measured using the commercially available ELISA assay.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Vahdat, MD, Principal Investigator — Study Principal Investigator
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No